CLINICAL TRIAL: NCT01617967
Title: A Phase 2, Open-Label, Multi-Dose, Dose Escalation Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous Infusions of ALN-TTR02 in Patients With TTR Amyloidosis
Brief Title: Safety and Tolerability of Patisiran (ALN-TTR02) in Transthyretin (TTR) Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTR02-002; 2012-000467-24 (EudraCT Number)
Expanded Access: NCT02939820 (Approved for marketing)
Record Dates: First submitted 2012-06-07; First posted 2012-06-13 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2018-10

CONDITIONS: TTR-mediated Amyloidosis
Keywords: RNAi therapeutic
MeSH Terms: interventions — patisiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Patisiran (ALN-TTR02) (Experimental): Two administrations of patisiran will be administered once every 4 weeks [Q4W]) in 4 sequential cohorts with escalating doses followed by optional cohorts with an alternative dosing regimen (once every 3 weeks [Q3W]), and an alternative premedication regimen.
  Interventions: Drug: Patisiran

INTERVENTIONS:
Drug: Patisiran — Participants received a single dose of patisiran as an intravenous (IV) infusion on Day 0 and Day 28 (Q4W). Optional cohorts received an alternative dosing regimen (once every 3 weeks [Q3W]: Day 0 and Day 21) and an alternative premedication regimen.
  Other Names: ALN-TTR02

SUMMARY:
This was a multiple dose, dose escalation study designed to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of patisiran (ALN-TTR02) in participants with transthyretin (TTR) mediated amyloidosis (ATTR).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index must be between 17 kg/m^2 and ≤ 33 kg/m^2;
* Women of child-bearing potential must have a negative pregnancy test, cannot be breast feeding, and must use appropriate contraception;
* Males agree to use appropriate contraception;
* Diagnosis of TTR amyloidosis;
* Adequate blood counts, liver and renal function;
* Willing to give written informed consent and are willing to comply with the study requirements.

Exclusion Criteria:

* Known human immunodeficiency virus (HIV) positive status or known or suspected systemic bacterial, viral, parasitic, or fungal infection;
* Received an investigational agent, other than tafamidis or diflunisal, within 30 days prior to first dose study drug administration;
* Prior liver transplant;
* Poor cardiac function;
* Considered unfit for the study by the Principal Investigator;
* Employee or family member of the sponsor or the clinical study site personnel.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (10):
- Clinical Trial Site, Boston, Massachusetts, United States
- Clinical Trial Site, Rio de Janeiro, Brazil
- France (2):
  - Clinical Trial Site, Le Kremlin-Bicêtre
  - Clinical Trial Site, Marseille
- Clinical Trial Site, Münster, Germany
- Portugal (2):
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- Spain (2):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Palma de Mallorca
- Clinical Trial Site, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Suhr OB, Coelho T, Buades J, Pouget J, Conceicao I, Berk J, Schmidt H, Waddington-Cruz M, Campistol JM, Bettencourt BR, Vaishnaw A, Gollob J, Adams D. Efficacy and safety of patisiran for familial amyloidotic polyneuropathy: a phase II multi-dose study. Orphanet J Rare Dis. 2015 Sep 4;10:109. doi: 10.1186/s13023-015-0326-6. PMID 26338094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 29 subjects were enrolled
Groups:
- Patisiran 0.010 mg/kg Q4W: Participants received 0.010 mg/kg of patisiran (ALN-TTR02) every four weeks (Q4W).
- Patisiran 0.050 mg/kg Q4W: Participants received 0.050 mg/kg of patisiran (ALN-TTR02) every four weeks.
- Patisiran 0.150 mg/kg Q4W: Participants received 0.150 mg/kg of patisiran (ALN-TTR02) every four weeks.
- Patisiran 0.300 mg/kg Q4W: Participants received 0.300 mg/kg of patisiran (ALN-TTR02) every four weeks.
- Patisiran 0.300 mg/kg Q3W: Participants received 0.300 mg/kg of patisiran (ALN-TTR02) every three weeks (Q3W).
- Patisiran 0.300 mg/kg Q3W Alternative: Participants received 0.300 mg/kg of patisiran (ALN-TTR02) every three weeks with alternative premedication regimen.
Period: Overall Study
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | Patisiran 0.300 mg/kg Q3W | Patisiran 0.300 mg/kg Q3W Alternative
Started | 4 | 3 | 3 | 7 | 3 | 9
Completed | 3 | 3 | 3 | 6 | 3 | 8
Not Completed | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Dosing Suspended by Sponsor | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | Patisiran 0.300 mg/kg Q3W | Patisiran 0.300 mg/kg Q3W Alternative | Total
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 3 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.96) | 55.7 (24.83) | 41.7 (2.52) | 58.7 (16.07) | 51.0 (16.09) | 54.7 (16.34) | 55.6 (15.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 4 | 1 | 2 | 9
  Male | 3 | 3 | 2 | 3 | 2 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 7 | 3 | 9 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Study Drug Discontinuation
Description: The number of participants experiencing at least one adverse event (AE), at least one serious adverse event (SAE) and study drug discontinuation (due to any reason).
Time Frame: Up to 56 days post first dose
Population: Intent-to-treat (ITT) population included all participants, who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | Patisiran 0.300 mg/kg Q3W | Patisiran 0.300 mg/kg Q3W Alternative
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 3 | 9
Participants
  At Least 1 AE | 1 | 3 | 2 | 7 | 3 | 7
  At Least 1 SAE | 0 | 0 | 0 | 1 | 0 | 1
  Study Drug Discontinuation For Any Reason | 1 | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Percentage Change From Baseline in Serum Transthyretin (TTR) Protein
Description: Percentage change of TTR relative to pretreatment/baseline levels is reported. For arms with a dosing regimen of Q4W TTR protein samples were measured on Days 28 and 56. For the arms with a dosing regimen of Q3W TTR protein samples were measured on Days 21 and 42.
Time Frame: Baseline to Day 21/28 and Day 42/56 depending on dosing regimen (Q3W/Q4W)
Population: ITT population included all participants, who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | Patisiran 0.300 mg/kg Q3W | Patisiran 0.300 mg/kg Q3W Alternative
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 3 | 8
Percentage
  Day 21 or 28 | -8.9 (9.91) | -21.7 (1.69) | -51.6 (22.84) | -73.9 (8.41) | -78.0 (7.55) | -80.7 (10.14)
  Day 42 or 56: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 8
  Day 42 or 56 | -20.3 (20.27) | -14.6 (15.8) | -44.7 (12.11) | -62.8 (25.11) | -78.7 (9.77) | -73.3 (19.55)

3. Secondary Outcome: Pharmacokinetic Parameters of Patisiran - Area Under the Concentration Curve From Time 0 to Last Measurable Time Point (AUC0-last)
Description: Pharmacokinetic profiles for patisiran (ALN-TTR02) were determined based on dosage and dosing frequency only, not premedication regimens. For arms with a dosing regimen of Q4W PK samples were taken on Days 0 and 28. For the arm with a dosing regimen of Q3W PK samples were taken on Days 0 and 21.
Time Frame: Predose, end of infusion and post-infusion at 5 minutes (min), 10 min, 30 min, 1 hour (h), 2 h, 4 h, 6 h, 24 h and 48 h on Day 0 and Day 21/28 depending on dosing regimen (Q3W/Q4W)
Population: The pharmacokinetic (PK) population included all participants, who received at least one dose of patisiran and had adequate data to determine a full pharmacokinetic profile. For PK outcome measures the two arms for patisiran 0.300 mg/kg at a dosing frequency of Q3W were combined and reported irrespective of premedication regimen.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- All Patisiran 0.300 mg/kg Q3W: All participants, who received 0.300 mg/kg of patisiran (ALN-TTR02) every three weeks irrespective of premedication regimen.
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | All Patisiran 0.300 mg/kg Q3W
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 12
ng*h/mL
  Day 0 | 2738 (3159) | 9604 (10588) | 18998 (5066) | 53724 (35814) | 39741 (33373)
  Day 21 or Day 28: number analyzed (Participants) | 3 | 3 | 3 | 6 | 11
  Day 21 or Day 28 | 2799 (2645) | 4884 (4652) | 27748 (17081) | 30013 (15935) | 25958 (28460)

4. Secondary Outcome: Pharmacokinetic Parameters of Patisiran - Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | All Patisiran 0.300 mg/kg Q3W
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 12
ng/mL
  Day 0 | 145 (23.4) | 672 (473) | 2560 (295) | 6053 (1326) | 4539 (1362)
  Day 21 or 28: number analyzed (Participants) | 3 | 3 | 3 | 6 | 11
  Day 21 or 28 | 106 (36.6) | 683 (391) | 3243 (986) | 3782 (1259) | 3314 (1253)

5. Secondary Outcome: Pharmacokinetic Parameters of Patisiran - Beta Elimination Half-life (t1/2 Beta)
Description: Pharmacokinetic profiles for patisiran were determined based on dosage and dosing frequency only, not premedication regimens. For arms with a dosing regimen of Q4W PK samples were taken on Days 0 and 28. For the arm with a dosing regimen of Q3W PK samples were taken on Days 0 and 21.
Time Frame: Predose, end of infusion and post-infusion at 5 minutes (min), 10 min, 30 min, 1 hour (h), 2 h, 4 h, 6 h, 24 h and 48 h on Day 0 and Day 21/28 depending on dosing frequency
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | All Patisiran 0.300 mg/kg Q3W
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 11
hour (h)
  Day 0: number analyzed (Participants) | 3 | 3 | 2 | 7 | 11
  Day 0 | 59.5 (59.3) | 39.6 (34.8) | 52.2 (NA) — Standard deviation not calculated for 2 participants | 48 (23.7) | 59.3 (17.2)
  Day 21 or 28: number analyzed (Participants) | 2 | 3 | 3 | 6 | 9
  Day 21 or 28 | 88.1 (NA) — Standard deviation not calculated for 2 participants | 39.4 (34.8) | 46.9 (6.05) | 50.2 (32.7) | 53.8 (15.2)

6. Secondary Outcome: Pharmacokinetic Parameters of Patisiran - Systemic Clearance (CL)
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | All Patisiran 0.300 mg/kg Q3W
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 11
L/h/kg
  Day 0: number analyzed (Participants) | 3 | 3 | 2 | 7 | 11
  Day 0 | 0.0163 (0.0248) | 0.123 (0.205) | 0.00883 (NA) — Standard deviation not calculated for 2 participants | 0.00851 (0.00606) | 0.0130 (0.0105)
  Day 21 or 28: number analyzed (Participants) | 3 | 3 | 3 | 6 | 11
  Day 21 or 28 | 0.0211 (0.0325) | 0.0844 (0.134) | 0.00658 (0.00324) | 0.0190 (0.0233) | 0.0222 (0.0138)

7. Secondary Outcome: Pharmacokinetic Parameters of Patisiran - Apparent Volume of Distribution at Steady State (Vss)
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | All Patisiran 0.300 mg/kg Q3W
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 11
L/kg
  Day 0: number analyzed (Participants) | 3 | 3 | 2 | 7 | 11
  Day 0 | 0.169 (0.092) | 0.279 (0.0896) | 0.428 (NA) — Standard deviation not calculated for 2 participants | 0.360 (0.197) | 0.588 (0.305)
  Day 21 or 28: number analyzed (Participants) | 2 | 2 | 3 | 5 | 9
  Day 21 or 28 | 0.264 (NA) — Standard deviation not calculated for 2 participants | 0.397 (NA) — Standard deviation not calculated for 2 participants | 0.305 (0.163) | 0.587 (0.251) | 0.881 (0.539)

8. Secondary Outcome: Pharmacokinetic Parameters of Patisiran - Renal Clearance (CLR)
Description: as for outcome 5
Time Frame: Predose (within 1 h of planned dosing start) and post-infusion at 0-6 h (pooled) on Day 0 and Day 21/28 depending on dosing frequency
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | All Patisiran 0.300 mg/kg Q3W
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 11
mL/h/kg
  Day 0 | 0.0153 (0.0307) | 0.0268 (0.0465) | 0.0129 (0.0223) | 0.0329 (0.0500) | 0.0334 (0.0631)
  Day 21 or 28: number analyzed (Participants) | 3 | 3 | 3 | 5 | 9
  Day 21 or 28 | 0.0320 (0.0555) | 0.253 (0.439) | 0.0410 (0.0710) | 0.0652 (0.0893) | 0.0563 (0.0979)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 56
Description: ITT population was the primary set for safety data and included all participants, who received at least 1 dose of study drug.
Arm/Group | Patisiran 0.010 mg/kg Q4W | Patisiran 0.050 mg/kg Q4W | Patisiran 0.150 mg/kg Q4W | Patisiran 0.300 mg/kg Q4W | Patisiran 0.300 mg/kg Q3W | Patisiran 0.300 mg/kg Q3W Alternative
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/7 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 1/7 | 0/3 | 1/9
Other Adverse Events (participants affected / at risk) | 1/4 | 3/3 | 2/3 | 7/7 | 3/3 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patisiran 0.010 mg/kg Q4W (N=4) | Patisiran 0.050 mg/kg Q4W (N=3) | Patisiran 0.150 mg/kg Q4W (N=3) | Patisiran 0.300 mg/kg Q4W (N=7) | Patisiran 0.300 mg/kg Q3W (N=3) | Patisiran 0.300 mg/kg Q3W Alternative (N=9)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patisiran 0.010 mg/kg Q4W (N=4) | Patisiran 0.050 mg/kg Q4W (N=3) | Patisiran 0.150 mg/kg Q4W (N=3) | Patisiran 0.300 mg/kg Q4W (N=7) | Patisiran 0.300 mg/kg Q3W (N=3) | Patisiran 0.300 mg/kg Q3W Alternative (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
Vessel puncture site haematoma (General disorders) | 0 | 1 | 2 | 2 | 1 | 1
Infusion related reaction (Immune system disorders) | 0 | 0 | 0 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2013-01-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT01617967/Prot_001.pdf
  • Statistical Analysis Plan (2013-07-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT01617967/SAP_000.pdf